CLINICAL TRIAL: NCT06047912
Title: Screening for Primary Aldosteronism in Hypertension With 24-hour URinary aLdosterone
Acronym: PURL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Ian B Wilkinson (Other)
Responsible Party: Sponsor-Investigator, Dr Ian B Wilkinson, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: A096651
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hypertension; Primary Aldosteronism; Urine Aldosterone
MeSH Terms: conditions — Hypertension; Hyperaldosteronism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study compares the positivity rates of two tests for screening for primary aldosteronism: plasma aldosterone renin ratio and 24-hour urine aldosterone in patients with young-onset hypertension with or without other clinical features of primary aldosteronism.

DETAILED DESCRIPTION:
Plasma aldosterone and renin measurements are subject to significant intra-individual variability, including variation related to posture, time of day and sodium balance. Aldosterone secretion is not constant and may be subject to diurnal variation. As such one-off testing of ARR, does not consider the salt status of the individual necessitating repetition of tests to ensure false negative or false positive test results are ruled out. The value of accumulated aldosterone in a 24-hour sample has the advantage that it does not depend on circadian variation. This pilot observational study will help establish the positivity rates of both standard plasma aldosterone renin ratio and 24-hour urine aldosterone, and the degree to which they correlate but will help establish if untargeted screening in young-onset hypertension is feasible and test the robustness of current standard guidelines for primary aldosteronism screening and case confirmation.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this trial only if all of the following criteria apply:

  * Aged 18 years and above.
  * Meets NICE criteria for a diagnosis of hypertension with an age of onset of hypertension between 18-60 years.
  * For cohort 2 (suspected primary aldosteronism): resistant hypertension, and/or hypertension with spontaneous or diuretic-induced hypokalaemia, and/or hypertension.

Exclusion Criteria:

* • Severe hypertension (sustained blood pressure of >200/110 mmHg) or a history of known secondary hypertension other than PA.

  * Contraindications to confirmatory testing with saline infusion or oral salt loading test as per standard clinical criteria such as known clinical diagnosis of heart failure, and/or chronic kidney disease stage 3b.
  * Known Pregnancy or breast feeding.
  * Lack of informed consent.
  * Any medical condition deemed unsuitable by investigator for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To enable the inclusion of a diverse population, representative of the UK in terms of ethnicity, and geographical and environmental factors that affect blood pressure and PA, we aim to conduct the study at several specialist hypertension sites in the UK. We will recruit patients referred to one of the study sites with hypertension (NICE definition) who fall into one of the following groups (cohorts):
  Cohort 1: Adult patients (18-75 years of age) with onset hypertension (≤60 years of age) but without other obvious features of PA Cohort 2: Adult patients (18-75 years of age) with onset hypertension (≤60 years of age) with one of the features: low serum potassium, or resistant hypertension.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Rates of positive and negative, Aldosterone renin ratio and 24-hr urine aldosterone in unselected patients with hypertension and in patients with suspected primary aldosteronism | 1 year
Degree of agreement between a positive/negative ARR and a positive/negative 24-hr urine aldosterone | 1 year

SECONDARY OUTCOMES:
Number of patients who required oral salt loading | 1 year
The predictive value of a positive aldosterone renin ratio or 24-hr urine aldosterone with a positive confirmatory test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, DM, MRCP, Study Chair — University of Cambridge
Locations (1):
- Vascular Research Clinic, Adenbrooke's Centre of Clinical Investigation, Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No